CLINICAL TRIAL: NCT07245251
Title: An Early-Phase Clinical Study Evaluating the Safety and Clinical Efficacy of STR-P004 in Subjects With Relapsed/Refractory CD19-Positive Acute Lymphoblastic Leukemia
Brief Title: To Evaluate the Safety, Tolerability, and Preliminary Antitumor Activity of STR-P004
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Starna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STR-P004-004
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphobkastic Leukemia
Keywords: STR-P004; ALL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose (Experimental): Five dose-escalation cohorts are planned within the dose range of AA mg/kg to BB mg/kg. The escalation follows a modified Fibonacci sequence
  Interventions: Drug: STR-P004

INTERVENTIONS:
Drug: STR-P004 — This study enrolls adult patients with B-cell acute lymphoblastic leukemia (B-ALL). Enrolled patients receive STR-P004 at the corresponding dose via intravenous infusion, administered four times

SUMMARY:
This is a single-arm, single-center, open-label, multiple-dose, dose-escalation early clinical study aimed at evaluating the safety, tolerability, pharmacokinetic characteristics, and preliminary antitumor activity of STR-P004 in subjects with relapsed/refractory CD19-positive acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
The study adopts a dose-escalation approach combining "accelerated titration" and "traditional 3+3" design. Five dose-escalation cohorts are planned within the dose range of AA mg/kg to BB mg/kg. The escalation follows a modified Fibonacci sequence (i.e., 2, 1.67, 1.5, 1.4, 1.33, 1.33… multiples), with faster escalation in the early stages to minimize patient exposure to ineffective doses and quickly reach the predicted effective dose range, followed by reduced escalation rates to ensure safety and explore efficacy.

ELIGIBILITY:
Inclusion Criteria:

Subjects with relapsed/refractory CD19-positive B-cell acute lymphoblastic leukemia who currently have poor prognosis treatment options:

1. Patients voluntarily sign the informed consent form;
2. Age between 18 and 65 years, regardless of gender;
3. Diagnosed with B-cell acute lymphoblastic leukemia and meeting any of the following conditions:

   * (1) Relapse: Relapse within 12 months after first remission following standard treatment;
   * (2) Refractory:

     1. No remission after ≥6 weeks of induction therapy or two courses of induction therapy;
     2. Relapse after ≥2 complete remissions (CR) or CR with incomplete hematologic recovery (CRi);
     3. First relapse after chemotherapy, with no remission after at least one salvage therapy;
   * d) Relapse after autologous or allogeneic hematopoietic stem cell transplantation;
4. Within 3 months before screening, bone marrow or peripheral blood tests show leukemia cells expressing CD19;
5. For Ph+ ALL patients, treatment failure with at least two tyrosine kinase inhibitors (TKIs) (including at least one second-generation TKI) or intolerance to TKI therapy; if the patient has a T315I mutation, TKI salvage therapy is not required;
6. During screening, the proportion of bone marrow blasts and immature lymphocytes is ≥5%;
7. Hemoglobin ≥60 g/L, platelets ≥30 × 10^9/L;
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
9. Adequate organ function, meeting the following criteria:

   * Aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN);
   * Alanine aminotransferase (ALT) ≤3 × ULN;
   * Total serum bilirubin ≤2 × ULN, unless combined with Gilbert's syndrome; patients with Gilbert's syndrome may be included if total serum bilirubin ≤3.0 × ULN and direct bilirubin ≤1.5 × ULN;
   * Serum creatinine ≤2.0 × ULN or creatinine clearance ≥60 mL/min (Cockcroft and Gault formula);
   * Minimum lung reserve: defined as ≤ grade 1 dyspnea and oxygen saturation >91% without oxygen supplementation;
   * International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (APTT) ≤1.5 × ULN;
10. Women of childbearing potential must have a negative blood/urine pregnancy test during screening and within 3 days before dosing. Any patient with reproductive potential must agree to use effective contraception throughout the study and for at least 2 years after the last dose of study treatment. As judged by the investigator, patients are considered to have reproductive potential if they are biologically capable of having children and have normal sexual activity. Female patients without reproductive potential (i.e., meeting at least one of the following criteria): hysterectomy, bilateral oophorectomy, bilateral tubal ligation, medically confirmed ovarian failure, or medically confirmed menopause (≥12 consecutive months of amenorrhea).

Exclusion Criteria:

Subjects meeting any of the following criteria cannot be enrolled:

1. Active central nervous system (CNS) leukemia (patients with CNS disease symptoms must undergo lumbar puncture to exclude CNS leukemia);
2. Isolated extramedullary relapse;
3. Prior CAR-T therapy or other genetically modified cell therapy within 6 months before screening;
4. Chemotherapy within 2 weeks before dosing, except for the following:

1.

* Pre-treatment chemotherapy as specified in the protocol;
* TKI and hydroxyurea must be discontinued 72 hours before cell infusion;
* 6-mercaptopurine, 6-thioguanine, methotrexate (standard dose), cytarabine (standard dose), vincristine, and asparaginase must be discontinued 1 week before cell infusion;
* Intrathecal chemotherapy for CNS leukemia prophylaxis must be discontinued 1 week before cell infusion; 2. Systemic corticosteroid therapy discontinued for less than 72 hours before dosing, except for physiological replacement doses (e.g., prednisone <10 mg/day or equivalent); 3. Acute graft-versus-host disease (GVHD) within 4 weeks before screening or moderate to severe chronic GVHD; systemic medication for GVHD within 4 weeks before dosing; 4. Active systemic autoimmune disease under treatment; 5. Any of the following:
* Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive;
* Hepatitis B e antibody (HBe-Ab) positive with HBV-DNA copy number above the lower limit of quantification;
* Hepatitis C antibody (HCV-Ab) positive;
* Anti-Treponema pallidum antibody (TP-Ab) positive;
* Human immunodeficiency virus (HIV) antibody positive;
* EBV-DNA or CMV-DNA copy number above the lower limit of quantification; 6. History or presence of other malignancies within 5 years before screening, except for those with low risk of recurrence as judged by the investigator after curative treatment and follow-up for more than 5 years; 7. Any of the following cardiac conditions:
* Left ventricular ejection fraction (LVEF) ≤45% (ECHO);
* New York Heart Association (NYHA) class III or IV congestive heart failure;
* Severe arrhythmia requiring treatment or clinically significant conduction abnormalities on ECG, including QTc interval ≥480 ms (QTcB = QT/RR^(1/2));
* Uncontrolled hypertension (systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg) or pulmonary hypertension despite standard treatment;
* Unstable angina;
* Myocardial infarction or coronary artery bypass graft/stent surgery within 6 months before dosing;
* Clinically significant valvular disease;
* Other cardiac diseases deemed unsuitable for enrollment by the investigator; 8. Clinically significant pleural effusion at screening; 9. History of epilepsy, cerebral ischemia/hemorrhage, cerebellar disease, or other active CNS diseases; 10. History of deep vein thrombosis or pulmonary embolism within 6 months before screening; 11. Known history of hypersensitivity to any component of the study drug; 12. Live vaccination within 6 weeks before screening; 13. Active infection at screening; 14. Expected lifespan less than 3 months; 15. Participation in another interventional clinical study within 3 months before screening involving investigational drugs not yet marketed, or within 5 half-lives for marketed drugs; or intention to participate in another clinical trial or receive anti-tumor therapy outside the protocol during the study; 16. Other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability endpoints | 12 months
  Dose-limiting toxicity (DLT), all adverse events (AEs)/serious adverse events (SAEs), and other safety evaluation indicators

IPD SHARING:
Plan to Share IPD: No